CLINICAL TRIAL: NCT05440344
Title: Pharmacokinetics of Imlunestrant in Participants With Hepatic Impairment
Brief Title: A Study of Imlunestrant (LY3484356) in Female Participants With Impaired Liver Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 18414; J2J-MC-JZLG (Other: Eli Lilly and Company)
Record Dates: First submitted 2022-06-27; First posted 2022-06-30 (Actual); Results first posted 2025-11-12 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-10

CONDITIONS: Hepatic Insufficiency; Healthy
MeSH Terms: conditions — Hepatic Insufficiency | interventions — Imlunestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Imlunestrant (Normal Hepatic Function) (Experimental): Participants received a single dose of Imlunestrant 400 milligrams (mg) administered orally on Day 1 in fasted state.
  Interventions: Drug: Imlunestrant
- Imlunestrant (Mild Hepatic Impairment) (Experimental): Participants received a single dose of Imlunestrant 400 mg administered orally on Day 1 in fasted state.
  Interventions: Drug: Imlunestrant
- Imlunestrant (Moderate Hepatic Impairment) (Experimental): Participants received a single dose of Imlunestrant 400 mg administered orally on Day 1 in fasted state.
  Interventions: Drug: Imlunestrant
- Imlunestrant (Severe Hepatic Impairment) (Experimental): Participants received a single dose of Imlunestrant 200 mg administered orally on Day 1 in fasted state.
  Interventions: Drug: Imlunestrant

INTERVENTIONS:
Drug: Imlunestrant — Administered orally.
  Other Names: LY3484356

SUMMARY:
The main purpose of this study is to measure how much of Imlunestrant (LY3484356) gets into the bloodstream and how long it takes the body to eliminate it in female participants with impaired liver function compared to female participants with normal liver function. The side effects and tolerability of Imlunestrant will also be evaluated. The study may last up to 46 days for each participant.

ELIGIBILITY:
Inclusion Criteria:

All Participants:

* Women not of childbearing potential may participate and include those who are infertile due to surgical sterilization (hysterectomy, bilateral oophorectomy, bilateral salpingectomy or tubal ligation), congenital anomaly such as mullerian agenesis; or postmenopausal
* Are between the body mass index (BMI) of 18.0 and 42.0 kilograms per meter squared (kg/m²), inclusive, at screening

Healthy Participants:

- Healthy females as determined by medical history, physical examination, and other screening procedures, with normal liver function

Participants with Impaired Liver Function:

* Females with chronic mild, moderate and severe liver impairment, assessed by Child-Pugh scoring
* Have diagnosis of chronic hepatic impairment (>6 months), with no clinically significant changes within 90 days prior to study drug administration.

Exclusion Criteria:

* Women of childbearing potential are excluded from the study.
* Have known allergies to imlunestrant or related compounds
* Have a history of alcoholism or drug/chemical abuse within 2 years prior to check-in
* Have received blood products within 2 months prior to check-in
* Have evidence of HIV infection and/or positive human HIV antibodies
* Have used or intend to use medications that are strong inhibiters or inducers of cytochrome P450 (CYP)3A4
* Who smoke more than 10 cigarettes or use the equivalent tobacco, smoking-cessation products, nicotine-containing products, or e-cigarettes (nicotine and non-nicotine) per day.
* Have a history or presence of cardiovascular (eg, symptomatic bradycardia with resting heart rate of <60 beats per minute), respiratory, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 27 (Actual)
Dates: Start 2022-07-05 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- United States (3):
  - Inland Empire Liver Foundation, Rialto, California
  - Orlando Clinical Research Center, Orlando, Florida
  - American Research Corporation at Texas Liver Institute, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study of Imlunestrant (LY3484356) in Female Participants With Impaired Liver Function — https://trials.lillytrialguide.com/en-US/trial/41FBumzAk7ebiIo0q9s7bX

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Imlunestrant (Normal Hepatic Function) | Imlunestrant (Mild Hepatic Impairment) | Imlunestrant (Moderate Hepatic Impairment) | Imlunestrant (Severe Hepatic Impairment)
Started | 9 | 6 | 6 | 6
Received at Least One Dose of Study Drug | 9 | 6 | 6 | 6
Completed | 9 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Imlunestrant (Normal Hepatic Function); Imlunestrant (Mild Hepatic Impairment); Imlunestrant (Moderate Hepatic Impairment): Participants received a single dose of Imlunestrant 400 mg administered orally on Day 1 in fasted state.
- Total: Total of all reporting groups
Arm/Group | Imlunestrant (Normal Hepatic Function) | Imlunestrant (Mild Hepatic Impairment) | Imlunestrant (Moderate Hepatic Impairment) | Imlunestrant (Severe Hepatic Impairment) | Total
Number analyzed (Participants) | 9 | 6 | 6 | 6 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (5.0) | 66.7 (3.1) | 59.2 (8.3) | 57.3 (3.1) | 60.8 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 6 | 6 | 27
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 3 | 3 | 15
  Not Hispanic or Latino | 5 | 1 | 3 | 3 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 1
  White | 8 | 6 | 5 | 6 | 25
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 | 6 | 6 | 6 | 27

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Maximum Observed Concentration (Cmax) of Imlunestrant
Description: PK: Cmax of Imlunestrant is reported.
Time Frame: Day 1 (Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144, 168, 192, 216, 240 hours post dose)
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Imlunestrant (Normal Hepatic Function) | Imlunestrant (Mild Hepatic Impairment) | Imlunestrant (Moderate Hepatic Impairment) | Imlunestrant (Severe Hepatic Impairment)
Number analyzed (Participants) | 9 | 6 | 6 | 6
nanograms per milliliter (ng/mL) | 58.0 (56) | 74.9 (47) | 87.6 (51) | 46.2 (49)

2. Primary Outcome: PK: Area Under the Concentration-time Curve From 0 to the Last Measurable Concentration (AUC[0-t]) of Imlunestrant
Description: AUC(0-t) of Imlunestrant is reported.
Time Frame: Day 1 (Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144, 168, 192, 216, 240 hours post dose)
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour per milliliter (ng*h/mL)
Groups:
- Imlunestrant (Severe Hepatic Impairment): Participants received a single dose of Pirtobrutinib 200 mg administered orally on Day 1 in fasted state.
Arm/Group | Imlunestrant (Normal Hepatic Function) | Imlunestrant (Mild Hepatic Impairment) | Imlunestrant (Moderate Hepatic Impairment) | Imlunestrant (Severe Hepatic Impairment)
Number analyzed (Participants) | 9 | 6 | 6 | 6
nanograms*hour per milliliter (ng*h/mL) | 1970 (51) | 2410 (27) | 4320 (50) | 2820 (47)

ADVERSE EVENTS:
Time Frame: Baseline up to 18 days
Description: All participants who received at least one dose of study drug.
Arm/Group | Imlunestrant (Normal Hepatic Function) | Imlunestrant (Mild Hepatic Impairment) | Imlunestrant (Moderate Hepatic Impairment) | Imlunestrant (Severe Hepatic Impairment)
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/6 | 1/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/9 | 0/6 | 2/6 | 2/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imlunestrant (Normal Hepatic Function) (N=9) | Imlunestrant (Mild Hepatic Impairment) (N=6) | Imlunestrant (Moderate Hepatic Impairment) (N=6) | Imlunestrant (Severe Hepatic Impairment) (N=6)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imlunestrant (Normal Hepatic Function) (N=9) | Imlunestrant (Mild Hepatic Impairment) (N=6) | Imlunestrant (Moderate Hepatic Impairment) (N=6) | Imlunestrant (Severe Hepatic Impairment) (N=6)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2023-12-18): https://cdn.clinicaltrials.gov/large-docs/44/NCT05440344/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-02): https://cdn.clinicaltrials.gov/large-docs/44/NCT05440344/SAP_001.pdf